CLINICAL TRIAL: NCT02074488
Title: Balancing Act: Impact on Falls in Older Adults With Vision Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maine (Other)
Collaborators: University of New England (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lenard W. Kaye, Director, UMaine Center on Aging; Professor, UMaine School of Social Work, University of Maine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21AG045661-01 (NIH); 1R21AG045661-01 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Postural Balance
Keywords: balance; gait

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fall Prevention Exercises (Experimental): Participant provided with Balancing Act exercise curriculum for completion at least fifteen minutes three times a week over a six month period.
  Interventions: Other: Balancing Act exercise curriculum; Other: Informational Brochure
- Informational brochure (Other): Participant receives an informational brochure and orientation to brochure contents.
  Interventions: Other: Informational Brochure

INTERVENTIONS:
Other: Balancing Act exercise curriculum — Balance improvement exercise curriculum titled "Balancing Act"
  Arms: Fall Prevention Exercises
Other: Informational Brochure — Informational Brochure on falls prevention

SUMMARY:
Falls are a significant issue for older adults with vision impairment. Medical conditions such as glaucoma and age-related macular degeneration that result in vision impairment negatively impact balance. Falling is 1.7 times more likely among older adults with vision impairment. In 2010 there were 9,146,026 older adults treated in emergency rooms for unintentional falls and injuries from falls are expected to cost the nation an estimated $54.9 billion dollars by 2020. Falls can lead to death, depression, and loss of independence. However, impaired balance is a modifiable risk factor for falls. A practical yet innovative falls prevention program has been developed that is designed to enhance balance and proprioception among older adults. This program, UExCEL (UNE-Exercise and Conditioning for Easier Living) Balancing Act, consists of simple exercises that can be done at home (15 minutes duration-3 times a week) during normal daily activities, requires only one brief training session, and no equipment. This study aims to establish an evidence base documenting the positive impact of Balancing Act exercises on balance and falls prevention for older adults with vision impairment. A randomized controlled trial of older adults with vision impairment (best corrected vision of 20/70 or worse) will be conducted over a 6-month period (control group n = 35 and Balancing Act intervention group n = 35) to determine the impact of Balancing Act on falls, fear of falling, pain, and activity levels. Factors that can be expected to affect its adoption and sustained use such as cost in the community and social support networks in the home will also be investigated. It is hypothesized that the Balancing Act intervention will decrease the number of falls experienced by older adults who have vision impairment by improving their gait and balance, reducing their fear of falling, increasing their physical activity, and reducing their pain.

The specific aims of the research are to: 1) Evaluate the impact of Balancing Act on standing balance control and proprioception for older adults who have vision impairment, using the Tinetti Gait & Balance Test, a validated tool for evaluating gait and balance and predicting fall risk; 2) Evaluate the impact of Balancing Act for older adults with vision impairment on falls, fear of falling, physical activity, and pain; and 3) Improve adherence to the Balancing Act exercise program by facilitating social networks. Data will be analyzed through: 1) a descriptive assessment of the baseline demographic characteristics of sample members, covariates, and outcome variables, as well as 2) a repeated measures design examining the impact of the intervention on study participants.

ELIGIBILITY:
Inclusion Criteria:

* 62 years or older
* Individual resides in his/her own home/apartment
* Best corrected vision of 20/70 or worse
* Is able to follow one step commands
* Individual is able to provide informed consent
* Individual can ambulate at least 200 feet (may use assistive devices)
* Score on Timed Get Up and Go test is equal to or greater than 12 seconds

Exclusion Criteria:

* Less than 62 years of age
* Individual does not reside in his/her own home/apartment
* Best corrected vision is better than 20/70
* Is not able to follow one step commands
* Is not able to provide informed consent
* Individual cannot ambulate at least 200 feet
* Score on Timed Get Up and Go test is less than 12 seconds

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Tinetti Gait and Balance Score at 6 months | 6 months

SECONDARY OUTCOMES:
Change from Baseline in Tinetti Gait and Balance Score at 4 months | 4 months

OTHER OUTCOMES:
Change from Baseline in Tinetti Gait and Balance Score at 2 months | 2 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of New England, Biddeford, Maine
  - University of Maine, Orono, Maine
  - The Iris Network, Portland, Maine